CLINICAL TRIAL: NCT00562016
Title: PROTECT II: A Prospective, Multi-center, Randomized Controlled Trial of the IMPELLA RECOVER LP 2.5 System Versus Intra Aortic Balloon Pump (IABP)in Patients Undergoing Non Emergent High Risk PCI
Brief Title: Protect II, A Prospective, Multicenter Randomized Controlled Trial
Acronym: PROTECT II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility on primary endpoint.Study confounded by statistically significant differences between the two arms re: atherectomy, duration of support.
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Carol Pekar/Director of Clinical and Regulatory Affairs, Abiomed Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7182007
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Artery Disease
Keywords: Patient undergoing scheduled PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMPELLA LP 2.5 (Experimental)
  Interventions: Device: IMPLELLA LP 2.5
- IABP Intra-aortic balloon pump (Active Comparator)
  Interventions: Device: IABP Intra-aortic balloon pump

INTERVENTIONS:
Device: IMPLELLA LP 2.5 — Insertion of the LP 2.5 IMPELLA circulatory support system that can be placed across the aortic valve using a single femoral site. The device pumps blood from the left ventricle into the ascending aorta at 2.5 L/min.
  Arms: IMPELLA LP 2.5
Device: IABP Intra-aortic balloon pump — IABP uses counterpulsation to provide 0.2L/min coronary flow
  Arms: IABP Intra-aortic balloon pump

SUMMARY:
The IMPELLA® 2.5 System will be superior to Intra Aortic Balloon Pump in preventing the composite rate of major adverse events during and after the PCI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Subject is indicated for a NON emergent percutaneous treatment of at least on de novo or restenotic lesion in a native coronary vessel or bypass graft.
* Patient presents with:

  * A compromised Ejection Fraction
  * Intervention on the last patent coronary conduit
  * Intervention on an unprotected left main artery or
  * Patient presenting with triple vessel disease.

Exclusion Criteria:

* ST elevation M.I.
* Pre procedure cardiac arrest within 24 hours.
* Subject in cardiogenic shock

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2007-10; Primary Completion 2011-04 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Composite rate of 10 major adverse events including death; MI;Stroke or TIA; and repeat revascularization. | 30 days +/- 10 days

SECONDARY OUTCOMES:
Maximum CPO decrease from baseline.Rate of in hospital major events compared between the IMPELLA and IABP. | In hospital events

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, Principal Investigator — Not affilicated with Abiomed
Locations (50):
- United States (44):
  - University of Alabama, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - California Cardiovascular/Washington Hospital, Fremont, California
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of Miami, Miami, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Medical College Of Georgia, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Massach General Hospital, Boston, Massachusetts
  - Brigham & Womens, Boston, Massachusetts
  - St. Elizabeths Medical Center, Boston, Massachusetts
  - Oakwood Hospital Wayne State University, Dearborn, Michigan
  - Henry Ford Medical, Detroit, Michigan
  - Harper Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Northern Michigan, Petoskey, Michigan
  - William Beaumont, Royal Oak, Michigan
  - Providence Hospital and Medical Centers, Southfield, Michigan
  - St. Louis University, St Louis, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Morristown Memorial, Morristown, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cardiovascular Research of Forsythe Medical, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist, Columbus, Ohio
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Veteran's Affairs Medical Center Dallas, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - University of Texas Medical School at Houston, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - St. Joseph's Hospital, Bellingham, Washington
  - University of Washington, Seattle, Washington
- Canada (5):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Royal Victoria Hospital at McGill, Montreal, Quebec
- Academic Medical Center, Amsterdam, Netherlands, Netherlands

REFERENCES:
- [Derived] Cohen MG, Matthews R, Maini B, Dixon S, Vetrovec G, Wohns D, Palacios I, Popma J, Ohman EM, Schreiber T, O'Neill WW. Percutaneous left ventricular assist device for high-risk percutaneous coronary interventions: Real-world versus clinical trial experience. Am Heart J. 2015 Nov;170(5):872-9. doi: 10.1016/j.ahj.2015.08.009. Epub 2015 Aug 15. PMID 26542494
- [Derived] Daubert MA, Massaro J, Liao L, Pershad A, Mulukutla S, Magnus Ohman E, Popma J, O'Neill WW, Douglas PS. High-risk percutaneous coronary intervention is associated with reverse left ventricular remodeling and improved outcomes in patients with coronary artery disease and reduced ejection fraction. Am Heart J. 2015 Sep;170(3):550-8. doi: 10.1016/j.ahj.2015.06.013. Epub 2015 Jun 26. PMID 26385039
- [Derived] Kovacic JC, Kini A, Banerjee S, Dangas G, Massaro J, Mehran R, Popma J, O'Neill WW, Sharma SK. Patients with 3-vessel coronary artery disease and impaired ventricular function undergoing PCI with Impella 2.5 hemodynamic support have improved 90-day outcomes compared to intra-aortic balloon pump: a sub-study of the PROTECT II trial. J Interv Cardiol. 2015 Feb;28(1):32-40. doi: 10.1111/joic.12166. PMID 25689546
- [Derived] Henriques JP, Ouweneel DM, Naidu SS, Palacios IF, Popma J, Ohman EM, O'Neill WW. Evaluating the learning curve in the prospective Randomized Clinical Trial of hemodynamic support with Impella 2.5 versus Intra-Aortic Balloon Pump in patients undergoing high-risk percutaneous coronary intervention: a prespecified subanalysis of the PROTECT II study. Am Heart J. 2014 Apr;167(4):472-479.e5. doi: 10.1016/j.ahj.2013.12.018. Epub 2014 Jan 3. PMID 24655695
- [Derived] Dangas GD, Kini AS, Sharma SK, Henriques JP, Claessen BE, Dixon SR, Massaro JM, Palacios I, Popma JJ, Ohman M, Stone GW, O'Neill WW. Impact of hemodynamic support with Impella 2.5 versus intra-aortic balloon pump on prognostically important clinical outcomes in patients undergoing high-risk percutaneous coronary intervention (from the PROTECT II randomized trial). Am J Cardiol. 2014 Jan 15;113(2):222-8. doi: 10.1016/j.amjcard.2013.09.008. PMID 24527505
- [Derived] O'Neill WW, Kleiman NS, Moses J, Henriques JP, Dixon S, Massaro J, Palacios I, Maini B, Mulukutla S, Dzavik V, Popma J, Douglas PS, Ohman M. A prospective, randomized clinical trial of hemodynamic support with Impella 2.5 versus intra-aortic balloon pump in patients undergoing high-risk percutaneous coronary intervention: the PROTECT II study. Circulation. 2012 Oct 2;126(14):1717-27. doi: 10.1161/CIRCULATIONAHA.112.098194. Epub 2012 Aug 30. PMID 22935569